CLINICAL TRIAL: NCT06427018
Title: Assessing the Expressions of Ezrin, Phosphorylated Ezrin, and Pip5k1α in the Airway Smooth Muscle of Asthmatic Patient
Brief Title: Expressions of Ezrin and Pip5k1α Proteins in Airway Smooth Muscle of Asthmatic Patients
Status: Recruiting | Type: Observational
Sponsor: Lei-Miao Yin (Other)
Collaborators: Yueyang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Shanghai 6th People's Hospital (Other); Xiangya Hospital of Central South University (Other); Baoshan Hospital, Shanghai University of Traditional Chinese Medicine (Unknown); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor-Investigator, Lei-Miao Yin, Prof., Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Other Study IDs: ShanghaiUTCM-0512
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Protein
Keywords: Asthma; Ezrin; Pip5k1α; Airway smooth muscle
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma group: No intervention.
  Interventions: Other: No intervention.
- Non-asthma group: No intervention.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Observational study with no intervention.

SUMMARY:
Asthma, a prevalent chronic respiratory affliction, significantly impinges upon the quality of life for affected individuals. Timely and appropriate diagnostic measures, coupled with efficacious therapeutic interventions, are paramount in mitigating exacerbations of symptoms and enhancing the life quality of patients.

Ezrin plays an important role in maintaining cell morphology, cell migration, cell adhesion and polarisation, but Ezrin expression in airway smooth muscle remains unclear.

Pip5k1α is an important kinase involved in intracellular phosphatidylinositol signalling pathways that may be involved in smooth muscle contraction and diastole.

Therefore, further studies are necessary to elucidate the changes of Ezrin and Pip5k1α in patients with asthma to provide a basis for investigating alternative treatments for asthma.

DETAILED DESCRIPTION:
Asthma is a complex and heterogeneous disease with a combination of genetic and environmental multifactors, which is mainly characterised by recurrent episodes of wheezing, shortness of breath, chest tightness and cough. The nature of the pathology manifests itself as a chronic inflammatory disease with abnormal antigen presentation and T-cell activation, and an imbalance of Th1/Th2 cells leading to dysfunction of airway smooth muscle cells. There is a lack of safe and effective medications against asthma for current treatment. For example, although glucocorticosteroids are the first-line drugs for asthma, only 12% of patients are able to use them in accordance with medical advice. β2 agonists are often used in combination with hormones, but up to 55% of asthmatics still fail to get effective control of their symptoms. Therefore, the development of innovative drugs with new targets and mechanisms has become the trend of asthma drug development at home and abroad. The discovery of new asthma targets will help to elucidate the asthma mechanism and solve a series of problems in clinical treatment.

Ezrin is one of the major members of the Ezrin-Radixin-Moesin (ERM) family, which plays an important role in the maintenance of cell morphology, cell migration, cell adhesion and polarisation. Pip5k1α is an important kinase involved in the intracellular phosphatidylinositol signaling pathway, which may be associated with the smooth muscle contraction and diastole related.

In a previous study, single-cell sequencing of lung tissue from asthmatic mice revealed that Ezrin and Pip5k1α were significantly increased in asthmatic airway smooth muscle cells. In vitro cellular experiments suggested that Ezrin and Pip5k1α inhibition could inhibit airway smooth muscle cell contraction, suggesting that inhibitors of both may provide a therapeutic advantage for reducing lung resistance in asthma. Therefore, further studies to elucidate the changes of Ezrin and Pip5k1α in asthma patients are warranted to provide a basis for the use of inhibitors of both as an alternative treatment for asthma.

ELIGIBILITY:
Inclusion Criteria:

* Lung tissue samples;
* The samples come from patients aged 18-70 years old, regardless of gender, who underwent lung tissue sampling for surgical indications during treatment;
* Paraffin sections of lung tissue from patients diagnosed with bronchial asthma, including tracheal smooth muscle;
* Paraffin sections of lung tissue from non-asthma patients, including tracheal smooth muscle.

Exclusion Criteria:

* Paraffin sections of lung tissue from patients who have been diagnosed with COPD;
* Other situations where the researcher deems it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referring to previous validation studies of target proteins in the literature, the sample size required for this validation experiment is related to multiple factors: (1) Selection of genes: mRNA differentially expressed genes will have a 50% probability of differential protein expression. (2) Antibody selection: Commercially available antibodies will be used for immunohistochemical detection of formalin-fixed, paraffin-embedded tissues with a success rate of up to 75%.
  According to previous validation studies of the target protein, the required samples are 60 in each group, for a total of 120 samples.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunofluorescence results | 6 months
  IF
Immunohistochemistry results | 6 months
  IHC

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Miao Yin, MD, Study Director — Yueyang Hospital, Shanghai University of Traditional Chinese medicine; Wei-Wei He, MD, Study Director — Shanghai 6th People's Hospital; Jun-Tao Feng, MD, Study Director — Xiangya Hospital of Central South University; Li Li, MD, Study Director — Baoshan Hospital, Shanghai University of Traditional Chinese Medicine; Xiao-Ling Xu, MD, Study Director — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Yueyang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.